CLINICAL TRIAL: NCT02529384
Title: Multiple B-value Diffusion-weighted Imaging in Evaluation of Breast Lesions：Compare Biexponential Model, Stretched Exponential Model, Conventional Monoexponential DWI and Pathological Specimens.
Brief Title: Multiple B-value Diffusion-weighted Imaging(DWI) in Evaluation of Breast Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDLL-2015128
Record Dates: First submitted 2015-06-16; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Breast Neoplasms; DWI
Keywords: Breast magnetic resonance imaging; Diffusion-weighted imaging; Multiple b-value diffusion weighted imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — After Surgical operation, specimen of lesion will be collected(Not every patient's specimen will be collected. We should be approved by patient themselves). For analyze the relation with biomarker from the MR imaging and pathological/molecular-biological biomarkers.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- malignant group: The lesion which is malignant tumors in breast
  Interventions: Other: Breast magnetic resonance scanning
- begin group: The lesion which is begin lesion in breast
  Interventions: Other: Breast magnetic resonance scanning
- The control group: Patient's ipsilateral or contralateral normal breast parenchyma were collected as a control group
  Interventions: Other: Breast magnetic resonance scanning

INTERVENTIONS:
Other: Breast magnetic resonance scanning — Just a muti-b value series in breast MRI

SUMMARY:
Breast cancer is the most commonly diagnosed cancer in women and its definite diagnose is still challenge for radiologist. This study is going to evaluate multi-b value diffusion weighted imaging in discrimination of breast benign and malignant lesions and explore the diagnostic effect of the combination of multi-parameter. At the same time, pathological specimens of patients will be collected. The relationship between magnetic resonance(MR) parameters and pathology biomarkers will be evaluated. Hope multi-b value diffusion weighted imaging can improve diagnosis for breast lesion and provide the basis for clinical treatment. The fundamental of pathology on MR signal change will be further expounded.

DETAILED DESCRIPTION:
Breast cancer is the most commonly diagnosed cancer in women and its definite diagnose is still challenge for radiologist. This study is going to evaluate multi-b values diffusion weighted imaging in discrimination of breast benign and malignant lesions and explore the diagnostic effect of the combination of multi-parameters. At the same time, pathological specimens of patients will be collected. The relationship between MR parameters and pathology biomarkers will be evaluated. By pre-contrast and post-contrast multi-b values diffusion weighted imaging series, patient's Apparent diffusion coefficient(ADC),tissue diffusivity (D), pseudo-diffusion coefficient (D*), perfusion fraction (f), distributed diffusion coefficient(DDC) and alpha will be evaluated. Parameters of benign , malignant breast lesions and ipsilateral or contralateral normal breast parenchyma as a control group will be measured. Receiver operating characteristic (ROC) curve analysis is used to test the ability of different parameters in differentiating malignant from begin lesions. After Surgical operation, specimen of lesion will be collected(Not every patient's specimen will be collected. The investigators should be approved by patient themselves). The biomarkers of specimen will be detected by pathological and molecular-biological methods.Then analyze the relation between parameters of the MR imaging and pathological/molecular-biological biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Female patient with breast lesion (Breast Imaging Reporting and Data System 2,3,4,5)
* Operation is take in Tang-du hospital

Exclusion Criteria:

* Postoperative patient
* Suffer radiotherapy,chemotherapy and endocrine treatment
* Serious image artifacts
* Lesion with diameter less than 3mm
* Scan during menstrual period
* Other magnetic resonance imaging contraindications

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with brest lesions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The values of Apparent diffusion coefficient (ADC, mm^2/s), tissue diffusivity (D, mm^2/s), pseudo-diffusion coefficient (D*, mm^ 2/s) measured from the DWI image | From first week to 92 week
  Parameters of multiple b-value and conventional DWI: ADC (mm^2/s), D (mm^2/s), D* (mm^2/s), distributed diffusion coefficient (DDC, mm^2/s).
The positive rates of molecular markers from the immunohistochemistry sections | From first week to 92 week
  Immunohistochemistry index (immunopositive rate, calculated with the numbers of positively labeled cells [2 fold increase vs the background] divided by the number of total cells) for estrogen receptor (ER), progesterone receptor(PR), Ki-67 (KI-67), Her 2 and Aquaporins.
The density measurement of microvessel density (MVD) and microlymphatic density (MLD) | From first week to 92 week
  MVD: the number of microvessels divided by the observing area; MLD: the number of lymphocytes divided by the observing area.

SECONDARY OUTCOMES:
Value of intraclass correlation coefficient (ICC) within inter-observe and intra-observe | From 92 week to 120 week.
  The intraclass correlation coefficient(ICC) of inter-observe and intra-observe.
The true-positive and true-negative rates for each parameter | From 92 week to 120 week.
  The true-positive, false-positve,true-negative and false negative rates for each paramter are first calculated. Then the diagonistic sensitivity and specificity of each parameter are decided.
The values of R and P for Pearson Correlation analyses between DWI parameters and molecular/morphological markers | From 120 week to 130 week.
  Correlation coefficient of each MR and pathological/molecular-biological biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Bao Ying Chen, M . D ., Study Director — Radiology department of Tang-Du hosipital
Locations (1):
- Tang-Du Hospital, Xi’an, Shanxi, China